CLINICAL TRIAL: NCT04125823
Title: Effects of Video Game-based Physical Activity Training in People With Multiple Sclerosis in the Inpatient Period During Relapse Treatment: a Pilot Randomized Controlled Trial
Brief Title: Video Game-based Physical Activity Training in People With Multiple Sclerosis During Relapse Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4992-GOA
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video game-based physical activity training (Experimental)
  Interventions: Behavioral: Video game-based physical activity training
- Conventional physiotherapy program (Active Comparator)
  Interventions: Behavioral: Conventional physiotherapy program

INTERVENTIONS:
Behavioral: Video game-based physical activity training — Based on the physical levels of the patients, appropriate games will be selected and video game based physical activity training will be started. Video games will be played with Xbox One with a motion sensor (Microsoft) and a 52'' Liquid Crystal Display. Depending on the prognosis of the patients, the grades and types of games will be changed.
  Sessions will be performed by a physiotherapist for 45 minutes once a day during the hospital stay.
  Arms: Video game-based physical activity training
Behavioral: Conventional physiotherapy program — A conventional physiotherapy program including balance, upper extremity, and core stabilization exercises will be implemented.
  Sessions will be performed by a physiotherapist for 45 minutes once a day during the hospital stay.
  Arms: Conventional physiotherapy program

SUMMARY:
The study aims to investigate the feasibility and acceptability of the video game-based physical activity training program in the inpatient period during relapse treatment. The secondary aims are to investigate its effectiveness on upper extremity functions, walking, balance, cognitive functions, quality of life, depression, and fatigue comparing to conventional rehabilitation in persons with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an inflammatory, demyelinating, neurodegenerative disease of the central nervous system. The most common clinical signs and symptoms are fatigue, spasticity, cognitive impairment, chronic pain, depression, decreased quality of life, and bladder and bowel dysfunction.

Current medical treatment is divided into three groups: disease-modifying, symptom management, and prognosis and relapse management. Intravenous methylprednisolone treatment is generally used in the management of relapses and prognosis. It is also thought that physiotherapy during the intravenous methylprednisolone treatment provides better treatment results. Therefore, treatment planning of people with MS during hospitalization should be done by a multidisciplinary team.

Studies have shown that video games based physical activity training as a non-pharmacological therapy may be an effective method for managing symptoms such as balance, gait, fatigue, and cognitive functions in people with MS, but its feasibility in the inpatient period is unknown.

The primary aim of the study is to investigate the feasibility and acceptability of the video game-based physical activity training program in the inpatient period. The secondary aims are to investigate its effectiveness on upper extremity functions, walking, balance, cognitive functions, quality of life, depression, and fatigue in persons with MS comparing to conventional rehabilitation.

Volunteers from people with MS who are in the inpatient period due to relapse in the Neurology Department, Faculty of Medicine, Dokuz Eylül University will participate in the study. In accordance with the inclusion criteria, 30 patients were randomly assigned to two groups: 15 patients in the game-based rehabilitation group and 15 patients in the conventional rehabilitation group. Based on the physical levels of the patients, appropriate games will be selected and video game based physical activity training will be started. Video games will be played with Xbox One with a motion sensor (Microsoft) and a 52'' Liquid Crystal Display. Depending on the prognosis of the patients, the grades and types of games will be changed. A conventional physiotherapy program including balance, upper extremity, and core stabilization exercises will be implemented. Treatments will be given by the physiotherapist for 45 minutes once daily during the hospital stay. Evaluations will be made before and after the treatment (discharge) and 4 weeks after the end of treatment. Physical and clinical evaluations will be made by physicians and physiotherapists, and cognitive evaluation will be performed by psychologists.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting or secondary progressive type of multiple sclerosis,
* Being able to walk at least 100 meters without resting,
* Being able to stably stand for half an hour,
* To be willing to participate in the study.

Exclusion Criteria:

* Having neurological disorder other than multiple sclerosis
* Orthopaedic surgery history covering the foot, ankle, knee, hip, or spine, affecting balance and walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment process: Number of people referred from physician and eligible for screening. Number of people attending interview with researcher. | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  Number of people referred from physician and eligible for screening. Number of people attending interview with researcher.
Acceptability - Prospective acceptability: Barriers (screening interview). | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  Barriers (screening interview). Burden (reasons for not taking part/discontinuation or dropping out).
Acceptability - Intervention coherence and adherence: Number of sessions attended. | Change from Baseline through Hospital Discharge, up to 10 days
  Number of sessions attended.
Acceptability - Experience (satisfaction, perceptions): Qualitative interview | Change from Baseline through Hospital Discharge, up to 10 days
  Qualitative interview (end of program).

SECONDARY OUTCOMES:
Timed 25-Foot Walk | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Timed 25-Foot Walk is a quantitative mobility and leg function performance test. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly and safely as possible. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score is the average time of the two completed trials. Higher time represents slower walking speed and more walking impairment.
12-Item Multiple Sclerosis Walking Scale | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The 12-Item Multiple Sclerosis Walking Scale is a patient-reported outcome measure that assesses the impact of multiple sclerosis on walking. It consists of 12 questions with Likert-type choose options concerning the limitations to walking due to multiple sclerosis during the past 2 weeks. The total score ranges 0 from 100. Higher scores indicate more impact of multiple sclerosis on walking.
Modified Fatigue Impact Scale | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Modified Fatigue Impact Scale provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The scale consists of 21 items with Likert-type choose options. The total score for the scale is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items. The total score ranges from 0 to 84. A higher score indicates higher level of fatigue.
2-Minute Walk Test | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The 2-Minute Walk Test is a submaximal exercise test that entails measurement of distance walked over a span of 2 minutes. The goal is for the individual to walk as far and fast as possible in 2 minutes. The total distance is recorded. Higher distance represents a better submaximal exercise capacity.
Six-Spot Step Test | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  Six-Spot Step Test reflects a complex array of sensorimotor functions, part of which are lower limb strength, spasticity, and coordination, as well as balance. The score is the average time of the four completed trials. Higher time represents more walking impairment.
Nine-Hole Peg Test | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Nine-Hole Peg Test is used to assess manual dexterity performance. It requires participants to repeatedly place and then remove nine pegs into nine holes, one at a time, as quickly as possible. Two trials for each hand are performed and the score is the average time. Higher scores indicate less manual dexterity performance.
Manual Ability Measure-36 | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Manual Ability Measurement-36 is a questionnaire on perceived ease or difficulty that a persons may experience when performing unilateral and bilateral activity of daily living tasks. During a semi-structured interview, the persons are asked to rate 36 unilateral and bilateral activity of daily living tasks using a 4-point scale. The score of the different tasks are summed up and transformed using a Rasch-derived conversion table. The Rasch-derived scores are ranged from 0 to 100. Higher scores indicate better manual ability.
Epworth Sleepiness Scale | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Multiple Sclerosis International Quality of Life Questionnaire | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Multiple Sclerosis International Quality of Life Questionnaire is a disease-specific, self-administered, multidimensional questionnaire, was co-developed and initially validated in 15 countries including Turkey. The questionnaire comprises 31 questions in 9 subscales: activities of daily living, psychological well-being, symptoms, relationships with friends, relationships with family, sentimental and sexual life, coping, rejection, and relationships with the healthcare system. All 9 dimensions and the index score were linearly transformed and standardized on a 0-100 scale, where 0 indicates the worst possible level of quality of life and 100 indicates the best level.
Hospital Anxiety and Depression Scale - Anxiety | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The scale aims to measure symptoms of generalized anxiety disorder and consists of 7 items. Each item is scored on a response-scale with four alternatives ranging between 0 and 3. Higher scores indicate higher symptoms.
Hospital Anxiety and Depression Scale - Depression | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The scale aims to measure symptoms of depression and consists of 7 items, seven items. Each item is scored on a response-scale with four alternatives ranging between 0 and 3. Higher scores indicate higher symptoms.
Symbol Digit Modalities Test | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Symbol Digit Modalities Test is used to assess information processing speed. Using a reference key, the test taker has 90 seconds to pair specific numbers with given geometric figures in the Symbol Digit Modalities Test. The correct matches are calculated as the test score. Higher scores indicate better information processing speed.
California Verbal Learning Test-II | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The California Verbal Learning Test-II is used to assess verbal memory. Higher scores indicate better verbal memory.
Revised Brief Visuospatial Memory Test | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Revised Brief Visuospatial Memory Test is used to assess visuospatial memory. Higher scores indicate better visuospatial memory.
Paced Auditory Serial Addition Test | Change from Baseline through Hospital Discharge, up to 10 days, and 4 weeks
  The Paced Auditory Serial Addition Test is used to assess auditory information processing speed and flexibility, as well as calculation ability. The score for the Paced Auditory Serial Addition Test is the total number correct out of 60 possible answers. Higher scores indicate higher cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Hospital, Neurology Department, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided